CLINICAL TRIAL: NCT05452525
Title: A Randomized, Open-label, Single Dose, 3-period, 6-treatment, Crossover Study to Compare the Pharmacokinetics and Safety/Tolerability of CKD-379 and Coadministration of D759, D745 and D150 in Healthy Subjects
Brief Title: Pharmacokinetics and Safety/Tolerability Profile of CKD-379
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A125_01BE2204
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: Test drug(CKD-379 I) Period 2: Test drug(CKD-379 II) Period 3: Reference drug(D759+D745+D150)
  Interventions: Drug: CKD-379 I; Drug: CKD-379 II; Drug: D759+D745+D150
- Sequence 2 (Experimental): Period 1: Test drug(CKD-379 I) Period 2: Reference drug(D759+D745+D150) Period 3: Test drug(CKD-379 II)
  Interventions: Drug: CKD-379 I; Drug: CKD-379 II; Drug: D759+D745+D150
- Sequence 3 (Experimental): Period 1: Test drug(CKD-379 II) Period 2: Reference drug(D759+D745+D150) Period 3: Test drug(CKD-379 I)
  Interventions: Drug: CKD-379 I; Drug: CKD-379 II; Drug: D759+D745+D150
- Sequence 4 (Experimental): Period 1: Test drug(CKD-379 II) Period 2: Test drug(CKD-379 I) Period 3: Reference drug(D759+D745+D150)
  Interventions: Drug: CKD-379 I; Drug: CKD-379 II; Drug: D759+D745+D150
- Sequence 5 (Experimental): Period 1: Reference drug(D759+D745+D150) Period 2: Test drug(CKD-379 I) Period 3: Test drug(CKD-379 II)
  Interventions: Drug: CKD-379 I; Drug: CKD-379 II; Drug: D759+D745+D150
- Sequence 6 (Experimental): Period 1: Reference drug(D759+D745+D150) Period 2: Test drug(CKD-379 II) Period 3: Test drug(CKD-379 I)
  Interventions: Drug: CKD-379 I; Drug: CKD-379 II; Drug: D759+D745+D150

INTERVENTIONS:
Drug: CKD-379 I — 1 tablet administration under fed condition
Drug: CKD-379 II — 1 tablet administration under fed condition
Drug: D759+D745+D150 — 3 tablet coadministration under fed condition

SUMMARY:
A study to compare the pharmacokinetics and safety/tolerability between CKD-379 tablet and D759, D745, D150 combination

DETAILED DESCRIPTION:
A randomized, open-label, single dose, 3-period, 6-treatment, crossover study to compare the pharmacokinetics and safety/tolerability of CKD-379 in healthy subjects under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Between 19 aged and 50 aged in healthy adult
* 50.0kg ≤ Body weight ≤ 90.0kg and 18.0kg/m2 ≤ body mass index (BMI) ≤ 27.0kg/m2

Exclusion Criteria:

* Have clinical significant medical history or disease that hepatobiliary system, kidney, nervous system, immune system, respiratory system, digestive system, urinary system, endocrine system(Type I or Type II Diabetes Mellitus, diabetic ketoacidosis ect.), hematological system, cardiovascular system(heart failure, Torsades de pointes etc.), mental illness
* Have clinical significant medical history or disease that urinary tract infection or genital infection including urosepsis, pyelonephritis
* Have a gastrointestinal disease(Crohn's disease, ulcer ect.) history that can effect drug absorption or surgery
* Those who are pregnant or breastfeeding
* Those who are deemed inappropriate to participate in clinical trial by investigators

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Cmax | 0~48hours
  Maximum plasma concentration of the drug
AUClast | 0~48hours
  Area under the concentration-time curve from the time of dosing to the last measurable concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jaeseong Oh, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No